CLINICAL TRIAL: NCT04096053
Title: 'Transgender Education for Affirmative and Competent HIV and Healthcare (TEACHH)': Protocol of Community-based Participatory Intervention Development and a Non-randomized Multi-site Pilot Study With Pre- Post-test Design
Brief Title: Transgender Education for Affirmative and Competent HIV and Healthcare
Acronym: TEACHH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Associate Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 00036238
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Stigma, Social; HIV/AIDS; Health Care Acceptability
MeSH Terms: conditions — Social Stigma; Acquired Immunodeficiency Syndrome; Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TEACHH (Experimental): The training workshop is designed as a 3-hour session for care providers. The training will be delivered by trans women. During this training, we plan to have providers: 1) discuss human rights for trans women; 2) teach providers about common words with which to discuss gender identity and expression, and develop a basic understanding of trans healthcare, HIV prevention, and HIV treatment, and how these types of healthcare affect trans women living with and affected by HIV; 3) discuss what it means to be trans-affirming in their work and how they can make their organizations more trans- affirming; and 4) have participants complete a case study to apply what they have learned to practice. These case studies will address issues affecting trans women who are immigrants/newcomers, trans women who are living with HIV, and trans women who experience other vulnerabilities.
  Interventions: Other: TEACHH

INTERVENTIONS:
Other: TEACHH — See arm/group description.

SUMMARY:
Educational workshops are an efficacious strategy to increase healthcare providers' ability to provide gender-affirming care for transgender (trans) people. This strategy may also reduce healthcare providers' stigma towards trans people and people living with HIV. There is less evidence, however, of educational workshops that address HIV prevention and care among trans women. This protocol details the development and pilot testing of the TEACHH: Transgender Education for Affirmative and Competent HIV and Healthcare intervention that aims to increase gender-affirming HIV care competency among healthcare providers.This community-based research (CBR) project involves intervention development and implementation of a non-randomized multi-site pilot study with pre- post-test design. First, the investigators will conduct a qualitative formative phase involving focus groups with 30 trans women and individual interviews with 12 providers to understand HIV care access barriers for trans women and elicit feedback on a proposed workshop. Second, the investigators will pilot test the intervention with 90-150 providers (n=30-50x3 in-person settings). Primary outcomes include feasibility (e.g., completion rate), workshop satisfaction, and willingness to attend another workshop. Secondary pre- and post-intervention outcomes, assessed directly preceding and following the workshop, include perceived competency, intention to provide gender-affirming HIV care, and attitudes/biases towards trans women with HIV. Primary outcomes will be summarized as frequencies and proportions (categorical variables) and means and standard deviations (continuous variables). The investigators will conduct paired-sample t tests to assess pre- and post-intervention differences for secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Workshop participants must be 18 years or older and identify as working at a location that provides health or social services to trans women or being in-training to work in health or social services (e.g., medical student, social work student). Workshop participants may include a mix of HIV- and non-HIV service providers.

Exclusion Criteria:

* Not fitting the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Workshop Recruitment Rate | 3 hours
  Number of people who participate in the workshop / Number of people invited to participate in the workshop
Workshop Completion Rate | 3 hours
  Number of people who finish all 3 hours of the workshop / Number of people who start the workshop
Survey completion rate | 3 hours
  Number of people who complete the post-survey/Number of people who complete the pre-survey
Satisfaction with the workshop | 3 hours
  Measured in two ways - satisfaction scale and willingness to attend another workshop on trans women with HIV

SECONDARY OUTCOMES:
attitudes/biases, perceived competency, and behavioral intention to provide gender- affirming HIV care to trans women living with HIV | 3 hours
  a scale adapted from (1) Nyblade et al.'s brief, standardized tool for measuring HIV- related stigma among health facility staff and (2) trans-specific questions from Bidell's Lesbian, Gay, Bisexual, and Transgender Development of Clinical Skills Scale (LGBT-DOCSS), an interdisciplinary self-assessment for health providers

CONTACTS AND LOCATIONS:
Locations (1):
- Factor-Inwentash Faculty of Social Work, University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacombe-Duncan A, Logie CH, Persad Y, Leblanc G, Nation K, Kia H, Scheim AI, Lyons T, Horemans C, Olawale R, Loutfy M. Implementation and evaluation of the 'Transgender Education for Affirmative and Competent HIV and Healthcare (TEACHH)' provider education pilot. BMC Med Educ. 2021 Nov 4;21(1):561. doi: 10.1186/s12909-021-02991-3. PMID 34732178
- [Derived] Lacombe-Duncan A, Logie CH, Persad Y, Leblanc G, Nation K, Kia H, Scheim AI, Lyons T, Loutfy M. 'Transgender Education for Affirmative and Competent HIV and Healthcare (TEACHH)': protocol of community-based intervention development and a non-randomised multisite pilot study with pre-post test design in Canada. BMJ Open. 2020 Jul 31;10(7):e034144. doi: 10.1136/bmjopen-2019-034144. PMID 32737085